CLINICAL TRIAL: NCT04317469
Title: Evaluation of Von Willebrand Factor as a Marker For Early Diagnosis of Acute Respiratory Distress Syndrome (A.R.D.S) in Comparison to Interleukin 6 [IL-6]
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia Elfawy, assistant professor of anesthiology and ICU , faculty of medicine , Ain Shams univeristy, Ain Shams University
Other Study IDs: research ethical comittee
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARDS group ,
  Interventions: Diagnostic Test: VWF measurement
- non ARDS group
  Interventions: Diagnostic Test: VWF measurement

INTERVENTIONS:
Diagnostic Test: VWF measurement — Plasma levels of both vWF and IL.6 were be measured on T=0 i.e. (at start of the study once the patient considered to be risky for A.R.D.S development to obtain their baseline levels), T=48 (after 48 hours), and T=72 (after 72 hours).
  Other Names: IL6 measurement

SUMMARY:
In this prospective study of 60patients, we tested the hypothesis That markedly elevated levels of plasma von Willebrand factor (VWF) a marker of endothelial cell injury might predict the development of acute respiratory distress syndrome (A.R.D.S) in risky patients. We compared our result to IL.6 as control biomarker for A.R.D.S development.

Acute lung injury was quantified on two -point scoring system (Berlin definition of ARDS and Murray score of acute lung injury).

Plasma levels of both vWF and IL.6 were be measured on T=0 i.e. (at start of the study once the patient considered to be risky for A.R.D.S development to obtain their baseline levels), T=48 (after 48 hours), and T=72 (after 72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years old of both sexes.
* risk factor for development of acute respiratory distress syndrome or acute lung injury either by:
* Direct lung injury includes: Severe pneumonia (infection), Breathing a vomited stomach contents (aspiration), Breathing harmful fumes or smoke, severe trauma to the chest or other accident that bruises the lungs.
* Indirect lung injury includes: sepsis, Severe injury or trauma with shock, blood transfusions , drug overdose acute pancreatitis, fracture of the long bones, near drowning ,anaphylaxis, uremia, fat embolus , and intracranial insult.

Exclusion Criteria:

* (1) pregnancy;
* (2) a preexisting medical condition with a life expectancy less than 3 months
* (3) evidence of cardiogenic pulmonary edema
* (4) age under 18 years old or above 80 years old
* (5) late stages of liver cell failure, renal failure
* (6) severe myocardial infarction
* (7) deep coma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients, admitted to the ICUs, staying >24 hrs will be randomly assigned to enter this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-03-21 (Estimated); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
level of vwf at 72 hours | 72 hours
  Plasma levels of both vWF and IL.6 were be measured on T=0 i.e. (at start of the study once the patient considered to be risky for A.R.D.S development to obtain their baseline levels), T=48 (after 48 hours), and T=72 (after 72 hours).